CLINICAL TRIAL: NCT05895877
Title: A Double-blind, Randomized, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Goofice® in Patients With Chronic Constipation
Brief Title: Evaluate the Efficacy and Safety of Goofice® (Elobixibat) in Patients With Chronic Constipation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Synmosa Biopharma Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYN-ELO-001
Record Dates: First submitted 2022-09-23; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2022-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goofice® (Active Comparator): Active ingredient:
  Elobixibat 5mg/tab
  Dosage and Frequency:
  Once daily before breakfast. The starting dose is total 10 mg of Goofice® (2 tablets). After 7 days of the start of the study treatment, the dosage may be adjusted according to symptoms among the dose levels of 5, 10, and 15 mg.However, the maximum daily dose is 15 mg (3 tablets).
  Interventions: Drug: Goofice®
- Goofice® Placebo (Placebo Comparator): Active ingredient/Excipients:
  The placebo drug is identical in appearance to the Goofice ® tablet with the same excipient ingredients, but without the active compound.
  Dosage and Frequency:
  Once daily before breakfast. The dosage and frequency is the same as active drug
  Interventions: Drug: Goofice® Placebo

INTERVENTIONS:
Drug: Goofice® — Once daily before breakfast.
  Arms: Goofice®
Drug: Goofice® Placebo — Once daily before breakfast.
  Arms: Goofice® Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial to evaluate the efficacy and safety of Goofice® in patients with chronic constipation.

DETAILED DESCRIPTION:
In order to enroll appropriate patients with chronic constipation, a 2-week constipation-related symptom intensity screening period will be established to investigate the number of bowel movements just prior to the study drug treatment initiation. Eligible subjects who fulfill all selection criteria for enrollment will be randomly assigned to receive Goofice® or placebo drug with 2:1 allocation ratio. The study drug will be received once daily approximately 30 minutes before breakfast in the 12-week treatment period. The starting dosing of Goofice® / placebo will be 10 mg (2 tablets) in treatment period. It is allowed to adjust the dosage among 5, 10, and 15 mg after 7 days after treatment initiation, if the dose adjusting criteria are met depending on symptoms. After treatment period, subjects will be followed up for 4 weeks to observe the effect of discontinuing treatment.

ELIGIBILITY:
Inclusion Criteria:

- At provisional enrollment

1. Men or women ≥ 20 years of age.
2. Include 2 or more of the following during the last 3 months with symptom onset of at least 6 months:

   1. Straining during more than 25% of bowel movements (BMs);)
   2. Lumpy or hard stools in 25% of BMs;
   3. Sensation of incomplete evacuation in more than 25% of all BMs;
   4. Sensation of anorectal blockage or obstruction in more than 25% of BMs;
   5. Manual maneuvers required in more than 25% of BMs;
   6. Fewer than 3 BMs per week.

      In addition to having at least 2 of the above criteria, the following must also apply:

   a. Loose stools are rarely present without the use of laxatives; b. Insufficient criteria for irritable bowel syndrome (IBS).
3. Ability to provide written consent. - At time of enrollment
4. A total of SBM frequencies < 6 times during the 2-week screening period.

Exclusion Criteria:

* At provisional enrollment

  1. Known or suspected allergy to components in elobixibat.
  2. Known or suspected organic constipation.
  3. Known or suspected symptomatic or drug-induced constipation.
  4. Known or suspected slow colon transit type constipation.
  5. Known or suspected excretory disorder constipation.
  6. Currently have or history of gastrointestinal obstruction.
  7. Currently have or history of abdominal hernia.
  8. History of laparotomy other than simple appendectomy.
  9. History of cholecystectomy or surgical or endoscopic intervention related to papillotomy.
  10. Subjects in whom the dosage regimens of medications, of which changing the dosage regimens is prohibited, will be changed after the day of informed consent.
  11. Cannot use the rescue medication (bisacodyl suppositories 10 mg).
  12. Pregnant, lactating or potentially pregnant women, women who wish to become pregnant from the time of the informed consent to the last observation/test point, or women who do not agree to use appropriate birth control methods. The acceptable effective contraception methods include: a. Male or female sterilization, implant, or intrauterine device; b. Injectable, pill, patch, ring plus one barrier method*; c. Two combined barrier methods*.

      * Effective barrier methods are diaphragm, male or female condoms, sponge, or spermicides (creams or gels that contain a chemical to kill sperm).
  13. Anemia, defined as hemoglobin ≤ 10 g/dL.
  14. Concurrent serious renal disease (creatinine ≥ 2.00 mg/dL) or liver disease (total bilirubin ≥ 3.0 mg/dL, or aspartate aminotransferase(AST) or alanine transaminase(ALT) ≥ 100 U/L).
  15. Concurrent clinical significant heart disease, including uncontrolled hypertension, arrhythmia, or heart failure.
  16. History of serious drug-induced allergy needs emergent medical intervention, such as anaphylaxis, angioedema, generalized urticaria or bronchospasm.
  17. Subjects have a history of cancer (other than basal cell or squamous cell carcinoma of the skin) unless the malignancy has been in a complete remission without maintenance chemotherapy for ≥ 5 years prior to the Screening visit.
  18. Subjects who are taking part in another clinical study, or subjects who take part in another clinical study within 12 weeks prior to the day of informed consent.
  19. Loss of weight greater than 5 kg one month before screening visit.
  20. Determined by the investigator to be not suitable for the conduct of the study for any other reasons.
  21. Subjects have a barium enema within 7 days of the Screening Visit.
* At time of enrollment

  22. Subjects have a clinically significant finding on colonoscopy performed as required in accordance with the American Gastroenterological Association (AGA) guidelines (within AGA time frames). If polyps are found and biopsied, pathology must be reviewed and must be negative for cancer before the subject may be enrolled in the study. 23. Used the rescue medication (bisacodyl suppositories 10 mg) at least 6 times during the 2-week screening period or subjects who used the rescue medication at least 3 times in Week -1 of the screening period. 24. Used the rescue medication for less than 72 hours after bowel movement during the 2-week screening period. 25. Mushy stool or watery stool (Bristol Stool Form Scale type 6 or 7) in SBM during the 2-week screening period. 26. Used prohibited medications/therapies during the 2-week screening period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Complete spontaneous bowel movement(CSBM) responder rate during 12 weeks treatment | 12 weeks
  * An overall CSBM responder is a subject who is a weekly CSBM responder for at least 9 of the 12 treatment weeks, including at least 3 of the last 4 treatment weeks.
  * A weekly CSBM responder will be defined as a subject with CSBM frequency of ≥ 3 times and CSBM frequency improved by ≥ 1 time from Week -1 of the screening period.
  * SBM is defined as defecation without laxative drug/enema or stool extraction. CSBM is defined as SBM without sensation of incomplete evacuation. In this study, when subjects used laxative drug at the day before initiation of screening period or rescue medication after initiation of screening period, defecation within 24 hours after the use of these medications will be not deemed as SBM or CSBM.

SECONDARY OUTCOMES:
Efficacy endpoint - Complete spontaneous bowel movement (CSBM) responder rate at Week 12 | 12 weeks
  - A responder will be defined as a subject with weekly (Week 12) CSBM frequency of ≥ 3 times and weekly (Week 12) CSBM frequency improved by ≥ 1 time from Week -1 of the screening period.
Efficacy endpoint - Spontaneous bowel movement (SBM) responder rate at Week 12 | 12 weeks
  - A responder will be defined as a subject with weekly (Week 12) SBM frequency of ≥3 times and weekly (Week 12) SBM frequency improved by ≥ 1 time from Week -1 of the screening period.
Efficacy endpoint - SBM and CSBM responder rate | 4 weeks
  - Changes of SBM and CSBM responder rate during follow-up period.
Efficacy endpoint - SBM frequency | 12 weeks
  - Changes in SBM frequency from screening period Week -1 at each week.
Efficacy endpoint - CSBM frequency | 12 weeks
  - Changes in CSBM frequency from screening period Week -1 at each week.
Efficacy endpoint - Mean stool consistency by Bristol Stool Form Scale | 12 weeks
  - The stool consistency is assessed based on the Bristol Stool Form Scale on a 7-grade scale.
  Grade / Interpretation
  1. / Separate hard lumps, like nuts (hard to pass)
  2. / Sausage shaped, but lumpy
  3. / Like a sausage, but with cracks on its surface
  4. / Like a sausage or snake, smooth and soft
  5. / Soft blobs with clear cut edges (passed easily)
  6. / Fluffy pieces with ragged edges, a mushy stool
  7. / Watery, no solid pieces, entirely liquid Mean stool consistency as measured at Week -1 and each treatment Week.
Exploratory endpoint - Patient Assessment of Constipation Quality of Life (PAC-QoL) | 12 weeks
  - Each item of the 28-item questionnaire (Appendix 1) is scored on a 5-point Likert-type scale from 0 to 4, with (0 = none/not at all, 1 = a little bit/a little bit of the time, 2 = moderately/some of the time, 3 = quite a bit/most of the time, 4 = extremely/all the time). Scores are reported overall and for each of the four subscales (physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction). An improvement (reduction) of ≥1 point in PAC-QoL score are considered clinically significant based on previous validation studies.
Exploratory endpoint - Patient Assessment of Constipation Symptoms (PAC-SYM) scores | 12 weeks
  - Symptom scores are evaluated using the PAC-SYM questionnaire, a validated, 12-item, Patient-reported outcome (PRO) instrument with abdominal, stool and rectal symptom subscales. Each item of the PAC-SYM is scored on a 5-point Likert-type scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe), with higher scores indicating greater symptom severity. An improvement (reduction) of ≥1 point in PAC-SYM score is considered clinically significant based on previous validation studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Clinical Trial Center, Taipei, Taiwan